CLINICAL TRIAL: NCT00870337
Title: Phase II Multicenter Study Evaluating the Tolerability and Efficacy of RAD001 (Everolimus) in Patients With Relapsed or Metastatic Endometrial Cancer
Brief Title: Everolimus in Treating Patients With Relapsed or Metastatic Endometrial Cancer
Acronym: ENDORAD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ARCAGY/ GINECO GROUP (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000633321; ARCAGY-ENDORAD; NOVARTIS-ARCAGY-ENDORAD; ARCAGY-GINECO-EN101; INCA-RECF0512; EUDRACT-2007-003002-10
Record Dates: First submitted 2009-03-26; First posted 2009-03-27 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Endometrial Cancer
Keywords: recurrent endometrial carcinoma; stage IV endometrial carcinoma; endometrial adenocarcinoma
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm (Experimental)
  Interventions: Drug: everolimus

INTERVENTIONS:
Drug: everolimus

SUMMARY:
RATIONALE: Everolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

PURPOSE: This phase II trial is studying how well everolimus works in treating patients with relapsed or metastatic endometrial cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Estimate the rate of non-progression after 3 months of treatment with everolimus in patients with relapsed or metastatic endometrial cancer.

Secondary

* Evaluate the partial and complete response rate after 3 months of treatment with everolimus in these patients.
* Evaluate the duration of response in these patients.
* Evaluate the clinical benefit after 6 months of treatment with everolimus in these patients.
* Evaluate the time to progression in these patients.
* Evaluate the progression-free and overall survival of these patients.
* Evaluate the nature, frequency, and severity of side effects of everolimus in these patients.

OUTLINE: This is a multicenter study.

Patients receive oral everolimus daily in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed monthly for 3 months and then every 3 months thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the endometrium

  * Metastatic disease after first- or second-line chemotherapy
* Previously treated with platinum-based therapy in the adjuvant or metastatic setting
* Must have ≥ 1 measurable metastatic lesion outside previously irradiated areas
* No locally recurrent resectable tumor
* No uncontrolled brain metastases

PATIENT CHARACTERISTICS:

* WHO performance status 0-1
* ANC ≥ 1,000/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9 g/dL
* Transaminases ≤ 2.5 times upper limit of normal (ULN) (≤ 5 times ULN in the presence of liver metastases)
* Alkaline phosphatase ≤ 2.5 times ULN
* Bilirubin ≤ 1.5 times ULN
* Creatinine clearance ≥ 50 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other cancer within the past 3 years except for curatively treated carcinoma in situ of the cervix or basal cell or squamous cell skin carcinoma
* No concurrent serious and/or uncontrolled disease that would preclude study participation, including any of the following:

  * Uncontrolled diabetes
  * Uncontrolled hypertension
  * Severe infection
  * Profound malnutrition
  * Unstable angina
  * NYHA class III-IV congestive heart failure
  * Ventricular arrhythmia
  * Coronary artery disease
  * Myocardial infarction within the past 6 months
  * Liver disease
  * Chronic renal failure
  * Progressive ulceration of the upper gastrointestinal tract
* No hypersensitivity to everolimus, sirolimus, or lactose
* No abnormalities ≥ grade 3
* No psychological, familial, social, or geographical reasons that would preclude study follow-up
* No history of poor compliance to medical treatment

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior experimental drugs (e.g., mTOR inhibitors)
* More than 21 days since prior and no other concurrent chemotherapy, hormonal therapy, or antitumor therapy
* More than 5 days since prior strong CYP3A4 inhibitors or inducers (e.g., rifabutin, rifampicin, clarithromycin, ketoconazole, itraconazole, voriconazole, ritonavir, or telithromycin)
* More than 30 days since other prior treatments
* No concurrent participation in another clinical trial that would interfere with the objectives of this study
* No concurrent anticoagulation, except for 1 mg of coumadin per day or low molecular weight heparin

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2008-03; Primary Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Rate of non-progression after 3 months of treatment with everolimus as assessed by RECIST criteria | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Laure Chauvenet, MD, Principal Investigator — Hotel Dieu de Paris
Locations (1):
- Hotel Dieu de Paris, Paris, France

REFERENCES:
- [Derived] Ray-Coquard I, Favier L, Weber B, Roemer-Becuwe C, Bougnoux P, Fabbro M, Floquet A, Joly F, Plantade A, Paraiso D, Pujade-Lauraine E. Everolimus as second- or third-line treatment of advanced endometrial cancer: ENDORAD, a phase II trial of GINECO. Br J Cancer. 2013 May 14;108(9):1771-7. doi: 10.1038/bjc.2013.183. Epub 2013 Apr 23. PMID 23612453
- [Derived] Tredan O, Treilleux I, Wang Q, Gane N, Pissaloux D, Bonnin N, Petit T, Cretin J, Bonichon-Lamichhane N, Priou F, Lavau-Denes S, Mari V, Freyer G, Lebrun D, Alexandre J, Ray-Coquard I. Predicting everolimus treatment efficacy in patients with advanced endometrial carcinoma: a GINECO group study. Target Oncol. 2013 Dec;8(4):243-51. doi: 10.1007/s11523-012-0242-9. Epub 2012 Dec 13. PMID 23238879